CLINICAL TRIAL: NCT02273817
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study Comparing the Bioquivalence of Ciclesonide Nasal Spray(Apotex Inc.) to That of Omnaris ™Nasal Spray (Sepracor, Inc.) in the Treatment of Seasonal Allergic Rhinitis
Brief Title: A Study Comparing The Bioequivalence Of Ciclesonide Nasal Spray (Apotex, Inc.) To That Of Omnaris™ Nasal Spray (Sepracor, Inc.) In The Treatment Of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apotex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CICE-NASU-05SB03-CE
Record Dates: First submitted 2014-10-14; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2012-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ciclesonide Nasal Spray (Apotex, Inc.) (Experimental): Ciclesonide nasal spray
  * Dosage form: contain the aqueous medium of each metered-dose pump spray formulation unit plus the active ingredient, ciclesonide.
  * Strength: 50 μg per actuation.
  * Batch/Lot number (Expiry date): JM6697 (May 2012)
  * Manufacturer: Apotex, Inc.
  Interventions: Drug: Ciclesonide nasal spray, 50 μg per actuation.
- Omnaris™ nasal spray (Active Comparator): Omnaris™ Nasal Spray,
  * Dosage form: contain the aqueous medium of each metered-dose pump spray formulation unit plus the active ingredient, ciclesonide
  * Strength: 50 μg per actuation
  * Batch/Lot number (Expiry date): 131657 (03/2012)
  * Manufacturer: Sepracor, Inc.
  Interventions: Drug: Ciclesonide nasal spray, 50 μg per actuation.
- Placebo (Placebo Comparator): Placebo
  * Dosage form: Contain the aqueous medium of each metered-dose pump spray formulation unit minus the active ingredient, ciclesonide.
  * Batch/Lot number (Expiry date): JR3808 (Nov 2012)
  * Manufacturer: Apotex, Inc.
  Interventions: Drug: Ciclesonide nasal spray, 50 μg per actuation.

INTERVENTIONS:
Drug: Ciclesonide nasal spray, 50 μg per actuation. — During placebo lead-in period: patients received placebo nasal spray, two actuations in each nostril once daily for 7 days.
  During treatment period: subjects were then assigned to one of the following three treatments according to the randomization scheme:
  1. Ciclesonide nasal spray: 50 μg per actuation, two actuations in each nostril once daily (200 μg per day) for 14 days.
  2. Omnaris™ nasal spray: 50 μg per actuation, two actuations in each nostril once daily (200 μg per day) for 14 days.
  3. Placebo nasal spray: 0 μg per actuation, two actuations in each nostril once daily for 14 days.

SUMMARY:
This study is to evaluate the equivalence of generic ciclesonide nasal spray with that of the marketed drug, Omnaris™ nasal spray, in the treatment of seasonal allergic rhinitis, and to evaluate the safety and tolerability of generic ciclesonide nasal spray compared with Omnaris™ nasal spray.

ELIGIBILITY:
Inclusion Criteria:

* If female of childbearing potential, is not pregnant (confirmed by negative urine pregnancy test) or lactating and must have used reliable birth control measures throughout the study.
* At least a 2-year reliable medical history consistent with SAR
* Positive skin test within 12 months of screening to at least one seasonal allergen present in the geographical area
* Capable of tolerating intranasal application of the IMP, willing and able to comply with the requirements of the protocol
* No clinically significant findings in physical and nasal examinations, and medical history.
* A reflective TNSS of at least 6 (out of 12) in the 24 hours prior to placebo lead-in visit.
* Successfully complete the placebo lead-in period.

Exclusion Criteria:

* - Signs or symptoms of nasal polyps, deviated septum, or any other condition which, in the opinion of the Investigator, could resulted in erroneous study data.
* Undergo nasal surgery or had nasal trauma within 3 months of screening.
* Active respiratory conditions or respiratory tract infection that require antibiotic treatment within 2 weeks of screening
* Persistent allergic rhinitis (PAR) that does not require or not expected to require active PAR treatment during the study period.
* Evidence of any unstable or clinically significant conditions that would place the subject at increased risk of complications, interfere with study participation, or confound any of the study objectives.
* Presence or history of clinically significant conditions which in the opinion of the Investigator would have compromised the safety of the subject or the conduct of the study.
* Use of corticosteroids, intranasal cromolyn, Leukotriene inhibitors, long or short acting antihistamines, intranasal or systemic decongestants prior to the start of the single-blind, placebo lead-in visit within the time periods specified in the protocol or receiving immunotherapy.
* Use of an investigational drug within 30 days before screening or during the study.
* Known or suspected hypersensitivity to corticosteroids.
* Inability to avoid exposure to chicken pox or measles.
* Infection requiring oral antibiotic treatment 2 weeks prior to screening.
* Previously identified as a placebo responder or known as a non responder to corticosteroids.
* History of alcohol, drug, or substance abuse in the 12 months prior to Visit 1 (screening).
* Positive for hepatitis B or C, or human immunodeficiency virus (HIV).
* Uncooperative or non compliant.
* Female subjects who planned to become pregnant during the conduct of the study.
* Current smoker (former smokers had to be 6 months smoke free).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Treatment Of Seasonal Allergic Rhinitis | 5 months
  Change from baseline in the combined reflective Total nasal symptom score (TNSS) (combined AM and PM reflective scores of runny nose, nasal congestion, nasal itchiness, and sneezing).

SECONDARY OUTCOMES:
Treatment Of Seasonal Allergic Rhinitis | 5 months
  Change from baseline in the combined AM and PM instantaneous scores of runny nose, nasal congestion, nasal itchiness, and sneezing.